CLINICAL TRIAL: NCT03614455
Title: An Open-label, Randomized, 2-period, 2-sequence Study to Evaluate the Single-dose Pharmacokinetics of Milademetan When Administered Alone or Concomitantly With Itraconazole or Posaconazole in Healthy Subjects
Brief Title: Pharmacokinetics (PK) Drug Interaction Study of Milademetan and Itraconazole or Posaconazole in Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: DS3032-A-U107
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — milademetan; Itraconazole; Cytochrome P-450 CYP3A Inhibitors; posaconazole

STUDY DESIGN:
Intervention Model Description: Prior to dosing on Day 1 of Treatment Period 1, subjects will be assigned to 1 of 2 sequences (sequences AB or AC), according to a pre-generated randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Milademetan alone (A) (Experimental): During Period 1, participants receive a single 100 mg milademetan oral dose on Study Day 1, with PK sampling to 168 hours post-dose (during the following 7-day washout period)
  Interventions: Drug: Milademetan
- Milademetan with itraconazole (AB) (Other): During Period 2, participants receive itraconazole, 200 mg twice daily (BID) on Study day 8 and 200 mg once daily (QD) on Study Days 9 through 20, along with a single 100 mg milademetan dose on Day 14
  Interventions: Drug: Milademetan; Drug: Itraconazole
- Milademetan with posaconazole (AC) (Other): During Period 2, participants receive 200 mg posaconazole three times daily (TID) on Study Days 8 through 20, along with a single 100 mg milademetan dose on Day 14
  Interventions: Drug: Milademetan; Drug: Posaconazole

INTERVENTIONS:
Drug: Milademetan — Milademetan 100 mg capsule for oral administration
  Other Names: Experimental product; DS-3032; CYP3A4 Substrate
Drug: Itraconazole — Itraconazole (200 mg) oral solution (20 mL of 10 mg/mL)
  Other Names: CYP3A4 Inhibitor
  Arms: Milademetan with itraconazole (AB)
Drug: Posaconazole — Posaconazole (200 mg) oral suspension (5 mL of 40 mg/mL)
  Other Names: CYP3A4 Inhibitor
  Arms: Milademetan with posaconazole (AC)

SUMMARY:
This will be an open-label, randomized, 3-treatment, 2-period, 2-sequence study in healthy subjects to evaluate the single-dose PK of milademetan when given as monotherapy and when administered with steady-state levels of the strong CYP3A4 inhibitors itraconazole or posaconazole.

The duration of the study for each individual subject will be approximately 49 days from the start of Screening through Study Discharge. Subjects will remain in-house for up to 23 days, including 22 overnight stays.

ELIGIBILITY:
Healthy participants with no clinically significant medical history or physical examination findings and who also meet all protocol-defined inclusion and exclusion criteria summarized as follows:

Inclusion Criteria:

* Has negative urine test for drugs of abuse, alcohol and tobacco
* If female, is surgically sterile or postmenopausal
* If male, agrees to protocol-defined contraceptive methods
* Has adequate hematologic, hepatic, and renal function as defined by the protocol
* Is able and willing to follow all study procedures
* Has provided a signed informed consent

Exclusion Criteria:

* Is female who is pregnant or breastfeeding
* Is unable to swallow oral medication
* Is unable to follow study procedures
* Has creatinine clearance < 90 mL/min at screening
* Is taking or has taken any medications or therapies outside of protocol-defined parameters
* Has history of or a known allergic reaction to azole antifungal agents
* Has any disease or condition that, per protocol or in the opinion of the investigator, might affect:

  1. safety and well-being of the participant or offspring
  2. safety of study staff

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of milademetan | pre-dose and then at 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC
Area under the plasma concentration-time curve extrapolated to infinity (AUCinf) of milademetan | within 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (Tmax) of milademetan | pre-dose and then at 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC
Area under the plasma concentration-time curve from time 0 to the time of last measurable concentration (AUC0-t) for milademetan | within 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC
Terminal elimination half-life (t½) of milademetan | within 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC
Apparent total body clearance (CL/F) of milademetan | within 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC
Apparent volume of distribution (Vz/F) | within 168 hours postdose
  Categories: alone (A), in sequence AB, in sequence AC

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/